CLINICAL TRIAL: NCT03825159
Title: A New Spinal Orthosis With an Integrated System of Electric Surface Stimulation and Heat Sensing for Adolescent Idiopathic Scoliosis
Brief Title: A New Spinal Orthosis for Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, physian, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCH-170102
Record Dates: First submitted 2018-12-30; First posted 2019-01-31 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES group (Experimental): Using spinal orthosis with an integrated system of electric surface stimulation and heat sensing.
  Interventions: Device: Spinal Orthosis with an Integrated System of Electric Surface Stimulation and Heat Sensing
- brace group (Active Comparator): Using spinal orthosis BRACE
  Interventions: Device: spinal orthosis

INTERVENTIONS:
Device: Spinal Orthosis with an Integrated System of Electric Surface Stimulation and Heat Sensing — The electrical stimulation technology integrated with the total contact spinal orthosis combines the external correction forces on the spinal skeleton from the passive orthosis with the muscle forces at the lateral trunk from the stimulation process.
  Arms: ES group
Device: spinal orthosis — The ventrally opened total contact spinal orthosis will be designed and made of Copolymer and Aliplast. Correcting pressure points have to use the pressure pads at relevant points.
  Other Names: Scoliosis brace
  Arms: brace group

SUMMARY:
The new device with digital technology provides a new avenue to enable clinicians to communicate wirelessly with the imbedded core system such that they can adjust the electrical stimulation parameters and retrieve the temperature data for further compliance analysis. The smart phone and cloud technology can be effectively applied for both security and convenience. The electrical stimulation technology integrated with the total contact spinal orthosis combines the external correction forces on the spinal skeleton from the passive orthosis with the muscle forces at the lateral trunk from the stimulation process. The electrical stimulation is purposely to tone the muscle in order to replace the external mechanical forces gradually. Ultimately, when being weaned off the orthosis, patients may maintain the correction.

DETAILED DESCRIPTION:
Spinal orthosis is an option to treat Adolescent Idiopathic Scoliosis (AIS) and is the most commonly used among conservative treatment. According to Scoliosis Research Society (SRS), orthotic treatment is indicated for AIS patients with curves greater than 25˚ but smaller than 45˚. However, the in-brace correction is hardly maintained and the effectiveness of orthotic treatment is limited, which has been an impetus to develop a more effective method for AIS patients to fulfill the unmet need. In order the orthosis is effective, biomechanical intervention and the patient compliance are two key factors. The purpose of this two-year project is to develop a new spinal orthosis in which an integrated system of electric surface stimulation and heat sensing is imbedded such that the AIS will be effectively treated with the mechanical orthosis plus a nocturnal use of electrical stimulation. In addition to the already stellar device, a totally new concept of spine erectability is proposed to provide evidence that can manifest the unique value of orthotic treatment as opposed to surgery. It is hypothesized that the new spinal orthosis would not only reduce the Cobb angle and apical rotation but also would strengthen the spine erectability in AIS patients. The new device with digital technology provides a new avenue to enable clinicians to communicate wirelessly with the imbedded core system such that they can adjust the electrical stimulation parameters and retrieve the temperature data for further compliance analysis. The smart phone and cloud technology can be effectively applied for both security and convenience. The electrical stimulation technology integrated with the total contact spinal orthosis combines the external correction forces on the spinal skeleton from the passive orthosis with the muscle forces at the lateral trunk from the stimulation process. The electrical stimulation is purposely to tone the muscle in order to replace the external mechanical forces gradually. Ultimately, when being weaned off the orthosis, patients may maintain the correction. With the spinal orthosis, the applied current in stimulation process would be reduced and the skin irritation would too. First year, there will be three tasks. An instrument will be developed for clinicians to assess the applicability of electrical surface stimulation to each AIS patient. System integration of the spinal orthosis with electrical surface stimulation and heat sensing will be accomplished. Clinical study of the effectiveness of passive spinal orthoses on 30 AIS subjects as a control group, where the Cobb angle, apical rotation and spine erectability will be measured before treatment and after. Second year, another 30 AIS patients will be recruited; the applicability of electrical surface stimulation will be assessed; and the new spinal orthosis will be applied to the experiment group. The Cobb angle, apical rotation and spine erectability will be measured before treatment and after for each subject. Independent t test will be carried out for the two groups to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* (1) the range of age should be from ten years old to seventeen years old and (2) the Cobb angle should be from 20°to 45°.

Exclusion Criteria:

* (1)not primary idiopathic scoliosis (2)Unable to wear the all-day brace

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Cobb angle | base line, 6th month and 12th month
  When measuring Cobb angle, the investigators should identify the upper and lower end vertebra. Then, the investigators draw perpendicular lines extending along the vertebral borders. The angle where two perpendicular lines meet is called Cobb angle
Change of Spine erectability | base line, 6th month and 12th month
  Spine erectability is to define the physiological ability of the spine to maintain it erect against gravity and will be assessed without wearing orthoses.
  The force F acting at the apex is the weights of the head and two upper limbs plus 7/17 trunk weight, which can be calculated with the readily available anthropometric data. The bending moment M at T8 equals the applied force F multiplies the lever arm d, which is the distance between the force and the weight line.
  SE=(Weight*7/17)*d/(Cobb angle in standing-Cobb angle in supine)
Change of Apical rotation | base line, 6th month and 12th month
  Apical rotation is the degree of apical vertebral rotation .The Raimondi method uses the projection of the vertebral pedicles and the width of the vertebra as a reference for the measuring. The largest axis of the pedicle is demarcated and measured on the side of the curve convexity, and the distance of the longitudinal line from the pedicle to the border of the vertebra on the convex side is measured. Those two values are transported to the ruler, and the value of the rotation is obtained.

SECONDARY OUTCOMES:
Back muscles surface ElectroMyoGraphy (EMG) | base line, 6th month and 12th month
  Use a non-invasive surface EMG tool to collect muscle activities on the upper and lower back area, while the subject performs the trunk flexion-extension-lateral rotation with standing posture.
Back movement pathway | base line, 6th month and 12th month
  Use cameras to record the back motion pathway during trunk flexion-extension & lateral rotations, while the subject performs the trunk flexion-extension-lateral rotation with standing posture.
Distributions of Pressure under the feet | base line, 6th month and 12th month
  Use a flat pressure mat embedded in the walkway to collect the foot pressure distribution during static standing and dynamic walking.
The nerve morphological connectivity | base line,12th month
  The subject's diffusion tensor features are extracted from functional Magnetic Resonance Imaging of head. The features would include the never connectivity, pathway, the size of nuclei.

CONTACTS AND LOCATIONS:
Overall Officials: TASEN WEI, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital Taiwan, Changhua, Taiwan